CLINICAL TRIAL: NCT00457275
Title: A Multicentre, Open-Label, Observational Local Study to Evaluate the LDL-C Lowering Effect of Ezetimibe as Prescribed in Daily Routine Practice in the South African Population
Brief Title: Observational Study to Evaluate LDL-C Lowering Effect of Ezetimibe (0653-070)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0653-070; 2007_012
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Duration of Therapy

INTERVENTIONS:
Drug: MK0653, ezetimibe / Duration of Treatment: 4 Weeks

SUMMARY:
To evaluate the LDL-C lowering in south african patients with primary hypercholesterolaemia after the addition of ezetimibe 10mg /day to ongoing therapy with a statin.

ELIGIBILITY:
Inclusion Criteria:

* Men or women >18 and <80 years of age
* Patients receiving statin therapy for a minimum period of 6 weeks prior to visit 1
* Female patients receiving hormone therapy (including hormone replacement therapy, any estrogen antagonist/agonist, or oral contraceptives) if maintained on a stable dose and regimen for at least 8 weeks prior to visit 1 and if willing to continue the same regimen throughout the study
* Liver enzyme levels less than or equal to 1.5 times the upper limit of normal with no active liver disease and CPK less than or equal to 1.5 times upper limit of normal at visit 1

Exclusion Criteria:

* Cardiovascular medications, such as beta-blockers, calcium-channel blockers,

angiotensin ii receptor antagonists or anticoagulants (i.e., warfarin) unless

treated with a stable regimen for at least 6 weeks prior to randomization and

patient agrees to remain on constant regimen for the duration of the study

* Patients on amiodarone hydrochloride will also be excluded
* General weight less than 50% of ideal body weight according to the 1983 metropolitan height and weight tables or weighing less than 100 lbs (45 kg)
* Hypersensitivity to HMG-COA reductase inhibitors
* Patient has congestive heart failure defined by nyha class III or IV, uncontrolled cardiac arrhythmias, unstable angina pectoris, or myocardial infarction; coronary artery bypass surgery, or angioplasty within 3 months of visit 1
* Taking lipid-lowering agents including fish oils, cholestin, bile-acid sequestrants

and niacin (grater than 200 mg/day) taken within 6 weeks and fibrates taken within 8 weeks prior to visit 1

* Taking medications that are potent inhibitors of cyp3a4, including cyclosporine,

systemic itraconazole or ketoconazole, erythromycin or clarithromycin,

nefazodone, verapamil and protease inhibitors

* Consumption of greater than 250 ml of grapefruit juice/day
* Taking oral corticosteroids unless used as replacement therapy for pituitary/adrenal disease and on a stable regimen for at least 6 weeks prior to visit 1
* Treatment with psyllium, other fiber-based laxatives, and/or OTC therapies

known to affect serum lipid levels, phytosterol margarines, unless treated with

a stable regimen for at least 6 weeks prior to visit 1 and patient agrees to remain on constant regimen for the duration of the study

* Women who are pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440
Dates: Start 2005-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Approval

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Raal F, Schamroth C, Patel J, Becker P. A multicentre, open-label, observational local study to evaluate the low-density lipoprotein cholesterol-lowering effect of ezetimibe as prescribed in daily routine practice in the South African population. Cardiovasc J Afr. 2007 Sep-Oct;18(5):325-9. PMID 17985033